CLINICAL TRIAL: NCT02403427
Title: The Voice Decision Support Expert System in Basal-bolus Insulin Therapy of Diabetes Patients.
Brief Title: The Expert System VoiceDiab in Children With Diabetes
Acronym: VoiceDiab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instytut Diabetologii Sp. z o.o. (Other)
Collaborators: Nalecz Institute of Biocybernetics and Biomedical Engineering, Polish Academy of Sciences (Other); National Center for Research and Development, Poland (Other)
Responsible Party: Principal Investigator, Ewa Pankowska, associate professor, Instytut Diabetologii Sp. z o.o.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PBS1/B9/13/2012-I
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Type 1 Diabetes Mellitus With Hyperglycemia; Type 1 Diabetes Mellitus With Hypoglycaemia
Keywords: Bolus calculator; Insulin pump; basal-bolus insulin therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VoiceDiab expert system (Experimental): the VoiceDiab system using before every main meal; three times per day.
  Interventions: Device: VoiceDiab expert system
- manual calculation (No Intervention): manula insulin calculation before every main meal; three times per day

INTERVENTIONS:
Device: VoiceDiab expert system — Decision support system VoiceDiab this is computer-based system constructed for mobile phone devices working on the server.
  Patients in experimental arm get the mobile phone application for 4 days. Glucose control will be done by two methods SMPG and CGM. Before every study's meal insulin dose with type of bolus will be indicate by VoiceDiab.
  Other Names: patient's decision supporting system
  Arms: VoiceDiab expert system

SUMMARY:
The purpose of this study to conduct the preliminary investigation on the efficacy and safety in terms of postprandial glucose value and the rates of hypoglycaemia when expert VoiceDiab system supports patient's decision on prandial insulin programming in insulin pump therapy.

DETAILED DESCRIPTION:
In children with type 1 diabetes glucose deterioration occurred every day and night leading into low satisfaction with treatment. Unstable glycemic profile resulting in high glycemic variability depends on the adjustment of insulin dosing to the current needs of the organism. The calculation of prandial insulin dosing is a complex process which involves such factors as preprandial blood glucose level, the amount of food taken, the glycemic index of carbohydrates, the insulin/carbohydrate exchange ratio, the active insulin level following the previous bolus. Currently, in patients treated with continuous subcutaneous insulin infusion (CSII) insulin pumps are equipped with bolus calculators which help to calculate prandial insulin dosing and thus contribute to improve post-prandial blood glucose levels.

The aim of the study was to determine whether the patient's support expert VoiceDiab system have stabilised diurnal glucose profile in children with type 1 diabetes treated with insulin pumps.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 1 diabetes at least 12 month prior screening visit
* Current treatment with basal-bolus regime and insulin pump for at least 12 weeks prior screening visit.
* HbAc < 11%
* Ability and willingness to adhere to the protocol including self-management and dealing with mobile device.

Exclusion Criteria:

* Multiply daily injection modality,
* Treatment with regular insulin,
* Use of any anti-diabetic agent,

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
postprandial glucose | 96 houres
  postprandial glucose with respect the hyperglycaemia above 180 mg/dl

SECONDARY OUTCOMES:
AUC | 240 mintues after each study's meal
  he Area Under The Curve (AUC) of postprandial glucose level over 240 minutes,
PPGE- postprandial glucose excursion | 96 houres
  Postprandial Glucose Excursions (PPGE), defined as the change in glucose concentration from before the meal to Peak Postprandial Glucose (PPG),
hypoglycemia | 96 houres
  Hypoglycaemic episodes over time of observation measeured by CGM
LBGI | 96 houres
  Low Blood Glucose Index ( LBGI) - as a one of the glucose variability parameters
Glucose variability parameters | 96 houres
  SD total (SDT)- from all days, SD within days (SDw); SD between time points (SDhh:mm); High Blood Glucose Index (HBGI)

OTHER OUTCOMES:
Quality of life | 10 days
  Patients well being when VoiceDiab system is implement
Patients' acceptances to use VoiceDiab system | 10 days
  based on the study's questioner

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Ladyzynski, PhD, Study Director — Institute of Biocybernetics and Biomedicin Engineering in Poland
Locations (1):
- Ewa Pankowska, Warsaw, Poland

REFERENCES:
- [Background] Pankowska E, Blazik M, Groele L. Does the fat-protein meal increase postprandial glucose level in type 1 diabetes patients on insulin pump: the conclusion of a randomized study. Diabetes Technol Ther. 2012 Jan;14(1):16-22. doi: 10.1089/dia.2011.0083. Epub 2011 Oct 20. PMID 22013887
- [Background] Blazik M, Pankowska E. The education of patients in prandial insulin dosing related to the structure of bolus calculators. Pediatr Endocrinol Diabetes Metab. 2010;16(4):301-5. PMID 21447273
- [Background] Kovatchev BP. Diabetes technology: markers, monitoring, assessment, and control of blood glucose fluctuations in diabetes. Scientifica (Cairo). 2012;2012:283821. doi: 10.6064/2012/283821. Epub 2012 Oct 17. PMID 24278682
- [Background] McCall AL, Cox DJ, Crean J, Gloster M, Kovatchev BP. A novel analytical method for assessing glucose variability: using CGMS in type 1 diabetes mellitus. Diabetes Technol Ther. 2006 Dec;8(6):644-53. doi: 10.1089/dia.2006.8.644. PMID 17109596
- [Result] Blazik M, Pankowska E. The effect of bolus and food calculator Diabetics on glucose variability in children with type 1 diabetes treated with insulin pump: the results of RCT. Pediatr Diabetes. 2012 Nov;13(7):534-9. doi: 10.1111/j.1399-5448.2012.00876.x. Epub 2012 May 14. PMID 22577884
- [Result] Pankowska E, Blazik M. Bolus calculator with nutrition database software, a new concept of prandial insulin programming for pump users. J Diabetes Sci Technol. 2010 May 1;4(3):571-6. doi: 10.1177/193229681000400310. PMID 20513322
- [Result] Pankowska E, Szypowska A, Lipka M, Szpotanska M, Blazik M, Groele L. Application of novel dual wave meal bolus and its impact on glycated hemoglobin A1c level in children with type 1 diabetes. Pediatr Diabetes. 2009 Aug;10(5):298-303. doi: 10.1111/j.1399-5448.2008.00471.x. Epub 2008 Oct 20. PMID 19175902
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed